CLINICAL TRIAL: NCT06666439
Title: LBC-Monitor: Liquid Biopsy Guided Tailoring of Therapy in Metastatic Lobular Breast Cancer (mILC): A Pilot Study of Longitudinal Tumor Burden Quantification Using Circulating Tumor DNA
Brief Title: Longitudinal Tumor Burden Quantification Using Circulating Tumor DNA in Metastatic Lobular Breast Cancer
Acronym: LBC-Monitor
Status: Recruiting | Type: Observational
Sponsor: Julia Foldi (Other)
Responsible Party: Sponsor-Investigator, Julia Foldi, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Other Study IDs: HCC 24-096
Record Dates: First submitted 2024-10-29; First posted 2024-10-30 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Invasive Lobular Carcinoma (mILC)
Keywords: CDK4/6 inhibitors (CDK4/6i); endocrine therapies (ET); estrogen and progesterone receptor (ER and PR) positive; human epidermal growth factor receptor 2 (HER2); ctDNA (circulating tumor DNA)
MeSH Terms: conditions — Carcinoma, Lobular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — circulating tumor DNA (ctDNA) - offers an alternative, minimally invasive approach for monitoring treatment response
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Diagnostic Test: circulating tumor DNA (ctDNA) — Signatera is based on a custom-designed multiplex polymerase chain reaction (mPCR) assay for each patient, targeting up to 16 mutations found in the patient's tumor during whole exome sequencing (WES) to create a unique tumor mutation signature.
  Other Names: Signatera

SUMMARY:
The goal of this study is to characterize early dynamic changes in ctDNA, which can aid in tailoring early therapy in patients with metastatic Invasive lobular carcinoma (ILC). Response assessment using ctDNA analysis could not only aid in de-escalation but also escalation strategies.

DETAILED DESCRIPTION:
Invasive lobular carcinoma (ILC) is the most common special histologic subtype of breast cancer (BC), comprising 10-15% of all invasive BCs and representing approximately 26,000-40,000 new cases annually in the United States. ILC has distinct morphological and biological features as well as clinical behavior compared to Invasive Ductal Carcinoma/breast carcinoma of no special type (NST). Given that most lobular breast cancers are ER+, in current clinical practice, newly diagnosed metastatic ILC (mILC) - either recurrent or de novo metastatic disease - is generally treated with sequential endocrine therapies (ET) until the tumor becomes endocrine resistant. ILC often presents as non-measurable disease on imaging, and it is often difficult to determine treatment response accurately using conventional imaging techniques. Therefore, novel ways of monitoring disease response are urgently needed. Analysis of circulating tumor DNA (ctDNA) offers an alternative, minimally invasive approach for monitoring treatment response, and can also identify molecular alterations that may predict resistance to endocrine therapies. Understanding early ctDNA dynamics during endocrine therapy is essential for future prospective clinical trials with adaptive molecularly driven designs. LBC-Monitor aims to define the optimal early timepoint of molecular response by ctDNA and the dynamics of these early changes as patients with mILC begin first line therapy with an antiestrogen agent such as an aromatase inhibitor or fulvestrant.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Patients must have histologically or cytologically confirmed invasive lobular breast cancer that is ER+ (> 1% staining) and HER2-negative as per ASCO/CAP guidelines with radiographical or clinical evidence of metastatic disease

   1. Lobular histology as assessed on either tissue collected from a metastatic lesion or from the patient's primary breast tumor (in case of recurrent metastatic disease)
   2. Patients with mixed ductal/lobular (NST/ILC) tumors are eligible to participate (with the ultimate goal to evaluate 20 patients with pure ILC)
   3. Patients must have tumor tissue available for whole exome sequencing for Signatera assay design
3. Prior therapies:

   1. Patients must not have received any therapy in the metastatic setting
   2. Patients could have received adjuvant therapy as indicated for their primary breast cancer
4. Age ≥ 18 years
5. Patients may be pre- or post-menopausal.

Exclusion Criteria:

1. Stage I-III breast cancer
2. Lack of lobular histology on tumor tissue biopsy
3. Other active cancer (previously treated cancer with no current evidence of disease is allowed)
4. ctDNA assay development is unattainable due to insufficient tumor tissue or sequencing failure

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients must have histologically or cytologically confirmed invasive lobular breast cancer that is ER+ (> 1% staining) and HER2-negative as per ASCO/CAP guidelines with radiographical or clinical evidence of metastatic disease, who plan to begin first line endocrine therapy with an aromatase inhibitor or fulvestrant alone for 12 weeks.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2029-10-31 (Estimated); Study Completion 2029-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in ctDNA | Baseline, at 4 weeks, at 8 weeks, at 12 weeks
  Change in circulating tumor DNA (ctDNA) is measured by MTM/ml in patients receiving first line endocrine therapy (an aromatase inhibitor or fulvestrant) for metastatic lobular breast cancer.

SECONDARY OUTCOMES:
Progression free survival (PFS) | Up to 2 years
  Length of time from start of treatment that patients live without disease progression per RECIST v1.1 in those with measurable disease on imaging. Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression). Data will be collected only in patients who completed the initial 12-week lead-in period with antiestrogen treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Foldi, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee Women's Hospital of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No